CLINICAL TRIAL: NCT01762319
Title: Cervical Ripening Before Endometrial Biopsy in Abnormal Uterine Bleeding (AUB) Using Sublingual Misoprostol 200 Mcg: A Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Cervical Ripening Before Endometrial Biopsy in Abnormal Uterine Bleeding Using Sublingual Misoprostol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIOGMVA002
Record Dates: First submitted 2012-12-11; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-09

CONDITIONS: Abnormal Uterine Bleeding Unrelated to Menstrual Cycle
MeSH Terms: interventions — Misoprostol; Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): 200 mcg Misoprostol SL 1 hour prior to fractional curettage
  Interventions: Drug: Misoprostol
- Vitamin B6 (Placebo Comparator): 100 mg Vitamin B6 SL 1 hr prior to fractional curettage
  Interventions: Drug: Vitamin B6

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Vitamin B6
  Other Names: Besix
  Arms: Vitamin B6

SUMMARY:
Abnormal uterine bleeding is common in Thai women. Fractional curettage is an diagnostic procedure of this condition. Traditionally, fractional curettage is performed under local anesthesia such as paracervical nerve block or intravenous meperidine.

Cervical dilatation using "metal cervical dilator" is a common method prior to perform fractional curettage. However, complication from this procedure can be occurred frequently, for example, uterine perforation, false tract formation and laceration of cervix.

Misoprostol is a prostaglandin E1 analogue which is commonly used in obstetrics and gynecology. Misoprostol transforms cervical component causing cervical ripening. This is very helpful for transcervical procedure because cervical dilatation is usually omitted. It can be prescribed in many route and sublingual route is the most effectiveness. Moreover, WHO supports the use of misoprostol in obstetrics and gynecology practice.

The hypothesis of this study is that "Misoprostol 200 micrograms sublingually is effective for cervical ripening before performing fractional curettage in patients with abnormal uterine bleeding" Double blind randomised controlled trial was performed using 26 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* thai women at the age over 35 years old
* presenting with abnormal uterine bleeding and have a plan to perform fractional curettage

Exclusion Criteria:

* uterine anomalies
* pregnancy
* pelvic inflammatory disease
* uncontrolled medical or psychological conditions
* known cases of gynecological diseases such as gynecological malignancies, abnormal pap smear
* Prostaglandin allergy
* Contraindicate to prostaglandin: asthma, mitral valve stenosis, glaucoma, sickle cell anemia

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
efficacy of 200 microgram Misoprostol for cervical ripening prior to performing fractional curettage in patients with abnormal uterine bleeding | 1 Year
  an efficacy of sublingual misoprostol in this study was dilatation of uterine cervix which was measured by a diameter of MVA cannula in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Korakot Sirimai, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Mittal S, Sehgal R, Aggarwal S, Aruna J, Bahadur A, Kumar G. Cervical priming with misoprostol before manual vacuum aspiration versus electric vacuum aspiration for first-trimester surgical abortion. Int J Gynaecol Obstet. 2011 Jan;112(1):34-9. doi: 10.1016/j.ijgo.2010.07.035. Epub 2010 Nov 26. PMID 21112054
- [Background] Allen R, O'Brien BM. Uses of misoprostol in obstetrics and gynecology. Rev Obstet Gynecol. 2009 Summer;2(3):159-68. PMID 19826573
- [Background] Cooper NA, Smith P, Khan KS, Clark TJ. Does cervical preparation before outpatient hysteroscopy reduce women's pain experience? A systematic review. BJOG. 2011 Oct;118(11):1292-301. doi: 10.1111/j.1471-0528.2011.03046.x. Epub 2011 Jul 29. PMID 21797959
- [Background] Saxena P, Salhan S, Sarda N. Role of sublingual misoprostol for cervical ripening prior to vacuum aspiration in first trimester interruption of pregnancy. Contraception. 2003 Mar;67(3):213-7. doi: 10.1016/s0010-7824(02)00517-6. PMID 12618256
- [Background] Saxena P, Salhan S, Sarda N. Sublingual versus vaginal route of misoprostol for cervical ripening prior to surgical termination of first trimester abortions. Eur J Obstet Gynecol Reprod Biol. 2006 Mar 1;125(1):109-13. doi: 10.1016/j.ejogrb.2005.07.022. Epub 2005 Sep 1. PMID 16139942
- [Background] Caliskan E, Filiz T, Yucesoy G, Coskun E, Vural B, Corakci A. Sublingual versus vaginal misoprostol for cervical ripening PRIOR TO manual vacuum aspiration under local anaesthesia: a randomized study. Eur J Contracept Reprod Health Care. 2007 Dec;12(4):372-7. doi: 10.1080/13625180701549758. PMID 17853158
- [Background] Saha SP, Bhattacharjee N, Baru G. Vaginal Misoprostol for Cervical Priming before Gynaecological Procedures on Non Pregnant Women. Int J Health Sci (Qassim). 2007 Jul;1(2):185-93. PMID 21475427
- [Background] Boonyarangkul A, Leksakulchai O. Comparison of level of pain between using manual vacuum aspiration and sharp curettage in management of abnormal uterine bleeding. J Med Assoc Thai. 2011 Dec;94 Suppl 7:S57-61. PMID 22619908
- [Background] Tansathit T, Chichareon S, Tocharoenvanich S, Dechsukhum C. Diagnostic evaluation of Karman endometrial aspiration in patients with abnormal uterine bleeding. J Obstet Gynaecol Res. 2005 Oct;31(5):480-5. doi: 10.1111/j.1447-0756.2005.00324.x. PMID 16176522